CLINICAL TRIAL: NCT00427193
Title: Comprehensive Assessment of Long-Term Effects of Reducing Intake of Energy (CALERIE)
Brief Title: CALERIE: Comprehensive Assessment of Long-Term Effects of Reducing Intake of Energy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00016876; PBRC U01-AG0204878; Tufts U01-AG020480; WashU U01-AG020487; DCRI/Duke U01-AG022132; AG0078
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Aging
Keywords: dietary restriction; disease /disorder prevention /control; nutrition of aging; bioenergetics; cardiovascular function; disease /disorder proneness /risk; insulin sensitivity / resistance
MeSH Terms: conditions — Disease Susceptibility; Insulin Resistance | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: all lab based assays were masked due to de-identified person and time interval measured. All physical measures were masked to intervention group status.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caloric Restriction (CR) (Experimental): 25% caloric restriction
  Interventions: Behavioral: Caloric Restriction (CR)
- Control, Ad libitum (AL) (Active Comparator): Ad libitum energy intake
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Caloric Restriction (CR) — Participants follow a diet with 25% fewer calories than calculated at baseline over a period of 24 months
  Arms: Caloric Restriction (CR)
Behavioral: Control — Participants continue their current diet for 24 months
  Arms: Control, Ad libitum (AL)

SUMMARY:
The purpose of this study is to test the hypothesis that two years of sustained 25% caloric restriction (CR) in men age 21-50 (inclusive) and women age 21-47 (inclusive) will slow aging and protect against age-related disease processes.

DETAILED DESCRIPTION:
The overall aim of CALERIE Phase 2 is to test the hypothesis that two years of sustained caloric restriction (CR), involving a reduction in energy intake to 75% of baseline (25% CR), in healthy, non-obese men aged 21-50 (inclusive) and women aged 21-47 (inclusive), will result in the same adaptive changes that were observed in a wide variety of animal studies. Particular emphasis is on the adaptive responses thought to be involved in slowing the aging process and protecting against age-related disease processes. Primary outcomes include core body temperature and resting metabolic rate. Secondary outcomes include risk factors for cardiovascular disease, inflammatory markers, immune function, psychological and physical function; oxidative changes in lipids, proteins, and DNA; and, risk factors for age-related conditions such as diabetes and body composition. An important secondary aim is to identify potential adverse effects of CR in humans.

The study will be conducted as a multi-center, parallel-group, randomized, controlled trial (RCT). A sample of 200 participants will be enrolled, and assigned to either the CR intervention or a control group. Control participants will be advised to simply continue their current diets. Participants in both treatment arms will be followed over a period of 24 months. A comprehensive set of evaluations will be performed prior to initiating the intervention, with follow-up evaluations at 1, 3, 6, 9, 12, 18 and 24 months afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Age must be between 21-50 (inclusive) for men and 21-47 (inclusive) for women
* Body mass index (BMI) must be greater than or equal to 22 and less than 28
* Female participants must use acceptable forms of contraception (barrier method, oral contraceptive, intra-uterine device, or similar) and be willing to continue using such a method while enrolled in the study

Exclusion Criteria:

* History or clinical manifestation of cardiovascular disease or an elevated blood pressure (greater than 140/90 mm Hg)
* Abnormal resting ECG
* History or clinical manifestation of diabetes
* History or clinical manifestation of cholelithiasis (the presence or formation of gallstones in the gallbladder or bile ducts)
* History of anaphylaxis, severe allergies, or asthma
* History or clinical manifestation of any other significant metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, immune, hepatic, renal, urologic disorders, or cancer that, in opinion of the investigator, would make the candidate ineligible for the study
* History of stomach or intestinal surgery (except appendectomy) or major abdominal, thoracic or non-peripheral vascular surgery within one year prior to the randomization date
* Any disease or condition that seriously affects body weight and/or body composition
* Potassium level above the upper limit of normal at the screening visit confirmed by a test repeated within two weeks
* Hemoglobin, hematocrit, RBC, or iron level below the lower limit of normal at the screening visit confirmed by a test repeated within two weeks
* Evidence of active liver disease or ALT levels above 1.5 times the upper limit of normal
* Practice a vegan dietary lifestyle
* History or clinical manifestation of any eating disorder
* Any history of pharmacologic treatment for a psychiatric disorder within one year prior to the randomization date or a history of more than one episode of a pharmacologic treatment for a psychiatric disorder within lifetime
* History of drug or alcohol abuse (up to 14 drinks a week are allowed) within the past two years
* BDI (Beck Depression Inventory) score of 20 or higher at screening or baseline
* Treatment with steroids for more than a month within five years prior to the randomization date, or short-term (less than a month) treatment with steroids within six months prior to the randomization date
* Regular use of other medications, except contraceptives
* Participated in the CALERIE Phase 1 studies
* Lost or gained 3 kg or more over the past six months
* A volunteer must be either a never-smoker of tobacco products or an ex-smoker who quit completely at least 12 months prior to the screening visit
* Donated blood within 30 days prior to the randomization date
* Concurrent participation in any other interventional study
* Breast-feeding or pregnant women or women intending to become pregnant before the scheduled end of the intervention
* Engaged in a regular program of physical fitness involving some kind of heavy physical activity (e.g., jogging, running or riding fast on a bicycle for 30 minutes or more) five or more times per week over the past year
* Unwilling to be assigned at random to the CR or control intervention
* Unwilling or unable to adhere to the rigors of the CR intervention over the entire two-year intervention period
* Unable or unwilling to discontinue dietary supplements or adhere to the alcohol consumption restrictions during the study
* Unwilling or unable to adhere to the rigors of the data collection and clinical evaluation schedule over the entire two-year period follow-up period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2007-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Kraus, MD, Principal Investigator — Duke Clinical Research Institute
Locations (3):
- United States (3):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Jean Mayer Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Result] Ravussin E, Redman LM, Rochon J, Das SK, Fontana L, Kraus WE, Romashkan S, Williamson DA, Meydani SN, Villareal DT, Smith SR, Stein RI, Scott TM, Stewart TM, Saltzman E, Klein S, Bhapkar M, Martin CK, Gilhooly CH, Holloszy JO, Hadley EC, Roberts SB; CALERIE Study Group. A 2-Year Randomized Controlled Trial of Human Caloric Restriction: Feasibility and Effects on Predictors of Health Span and Longevity. J Gerontol A Biol Sci Med Sci. 2015 Sep;70(9):1097-104. doi: 10.1093/gerona/glv057. Epub 2015 Jul 17. PMID 26187233
- [Result] Rochon J, Bales CW, Ravussin E, Redman LM, Holloszy JO, Racette SB, Roberts SB, Das SK, Romashkan S, Galan KM, Hadley EC, Kraus WE; CALERIE Study Group. Design and conduct of the CALERIE study: comprehensive assessment of the long-term effects of reducing intake of energy. J Gerontol A Biol Sci Med Sci. 2011 Jan;66(1):97-108. doi: 10.1093/gerona/glq168. Epub 2010 Oct 5. PMID 20923909
- [Result] Racette SB, Rochon J, Uhrich ML, Villareal DT, DAS SK, Fontana L, Bhapkar M, Martin CK, Redman LM, Fuss PJ, Roberts SB, Kraus WE. Effects of Two Years of Calorie Restriction on Aerobic Capacity and Muscle Strength. Med Sci Sports Exerc. 2017 Nov;49(11):2240-2249. doi: 10.1249/MSS.0000000000001353. PMID 29045325
- [Result] Belsky DW, Huffman KM, Pieper CF, Shalev I, Kraus WE. Change in the Rate of Biological Aging in Response to Caloric Restriction: CALERIE Biobank Analysis. J Gerontol A Biol Sci Med Sci. 2017 Dec 12;73(1):4-10. doi: 10.1093/gerona/glx096. PMID 28531269
- [Result] Martin CK, Bhapkar M, Pittas AG, Pieper CF, Das SK, Williamson DA, Scott T, Redman LM, Stein R, Gilhooly CH, Stewart T, Robinson L, Roberts SB; Comprehensive Assessment of Long-term Effects of Reducing Intake of Energy (CALERIE) Phase 2 Study Group. Effect of Calorie Restriction on Mood, Quality of Life, Sleep, and Sexual Function in Healthy Nonobese Adults: The CALERIE 2 Randomized Clinical Trial. JAMA Intern Med. 2016 Jun 1;176(6):743-52. doi: 10.1001/jamainternmed.2016.1189. PMID 27136347
- [Derived] Racette SB, Silver RE, Barry VG, DeGraff JJ, Gunning JA, Kebbe M, Gilhooly CH, Das SK. Diet quality and nutritional adequacy during a 2-year calorie restriction intervention: the Comprehensive Assessment of Long-Term Effects of Reducing Intake of Energy 2 trial. Am J Clin Nutr. 2025 Dec 29;123(3):101182. doi: 10.1016/j.ajcnut.2025.101182. Online ahead of print. PMID 41475553
- [Derived] Ryan CP, Corcoran DL, Banskota N, Eckstein Indik C, Floratos A, Friedman R, Kobor MS, Kraus VB, Kraus WE, MacIsaac JL, Orenduff MC, Pieper CF, White JP, Ferrucci L, Horvath S, Huffman KM, Belsky DW. The CALERIE Genomic Data Resource. Nat Aging. 2025 Feb;5(2):320-331. doi: 10.1038/s43587-024-00775-0. Epub 2024 Dec 13. PMID 39672986
- [Derived] Glasbrenner C, Hochsmann C, Pieper CF, Wasserfurth P, Dorling JL, Martin CK, Redman LM, Koehler K. Prediction of individual weight loss using supervised learning: findings from the CALERIETM 2 study. Am J Clin Nutr. 2024 Nov;120(5):1233-1244. doi: 10.1016/j.ajcnut.2024.09.003. Epub 2024 Sep 11. PMID 39270937
- [Derived] Ryu S, Spadaro O, Sidorov S, Lee AH, Caprio S, Morrison C, Smith SR, Ravussin E, Shchukina I, Artyomov MN, Youm YH, Dixit VD. Reduction of SPARC protects mice against NLRP3 inflammasome activation and obesity. J Clin Invest. 2023 Oct 2;133(19):e169173. doi: 10.1172/JCI169173. PMID 37781916
- [Derived] Silver RE, Roberts SB, Kramer AF, Chui KKH, Das SK. No Effect of Calorie Restriction or Dietary Patterns on Spatial Working Memory During a 2-Year Intervention: A Secondary Analysis of the CALERIE Trial. J Nutr. 2023 Mar;153(3):733-740. doi: 10.1016/j.tjnut.2023.01.019. Epub 2023 Jan 14. PMID 36805108
- [Derived] Dorling JL, Ravussin E, Redman LM, Bhapkar M, Huffman KM, Racette SB, Das SK, Apolzan JW, Kraus WE, Hochsmann C, Martin CK; CALERIE Phase 2 Study Group. Effect of 2 years of calorie restriction on liver biomarkers: results from the CALERIE phase 2 randomized controlled trial. Eur J Nutr. 2021 Apr;60(3):1633-1643. doi: 10.1007/s00394-020-02361-7. Epub 2020 Aug 14. PMID 32803412
- [Derived] Thomas DM, Clark N, Turner D, Siu C, Halliday TM, Hannon BA, Kahathuduwa CN, Kroeger CM, Zoh R, Allison DB. Best (but oft-forgotten) practices: identifying and accounting for regression to the mean in nutrition and obesity research. Am J Clin Nutr. 2020 Feb 1;111(2):256-265. doi: 10.1093/ajcn/nqz196. PMID 31552422
- [Derived] Dorling JL, Bhapkar M, Das SK, Racette SB, Apolzan JW, Fearnbach SN, Redman LM, Myers CA, Stewart TM, Martin CK; CALERIE Study Group. Change in self-efficacy, eating behaviors and food cravings during two years of calorie restriction in humans without obesity. Appetite. 2019 Dec 1;143:104397. doi: 10.1016/j.appet.2019.104397. Epub 2019 Aug 6. PMID 31398376
- [Derived] Kraus WE, Bhapkar M, Huffman KM, Pieper CF, Krupa Das S, Redman LM, Villareal DT, Rochon J, Roberts SB, Ravussin E, Holloszy JO, Fontana L; CALERIE Investigators. 2 years of calorie restriction and cardiometabolic risk (CALERIE): exploratory outcomes of a multicentre, phase 2, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Sep;7(9):673-683. doi: 10.1016/S2213-8587(19)30151-2. Epub 2019 Jul 11. PMID 31303390
- [Derived] Broskey NT, Marlatt KL, Most J, Erickson ML, Irving BA, Redman LM. The Panacea of Human Aging: Calorie Restriction Versus Exercise. Exerc Sport Sci Rev. 2019 Jul;47(3):169-175. doi: 10.1249/JES.0000000000000193. PMID 30998529
- [Derived] Guo J, Brager DC, Hall KD. Simulating long-term human weight-loss dynamics in response to calorie restriction. Am J Clin Nutr. 2018 Apr 1;107(4):558-565. doi: 10.1093/ajcn/nqx080. PMID 29635495
- [Derived] Redman LM, Smith SR, Burton JH, Martin CK, Il'yasova D, Ravussin E. Metabolic Slowing and Reduced Oxidative Damage with Sustained Caloric Restriction Support the Rate of Living and Oxidative Damage Theories of Aging. Cell Metab. 2018 Apr 3;27(4):805-815.e4. doi: 10.1016/j.cmet.2018.02.019. Epub 2018 Mar 22. PMID 29576535
- [Derived] Das SK, Roberts SB, Bhapkar MV, Villareal DT, Fontana L, Martin CK, Racette SB, Fuss PJ, Kraus WE, Wong WW, Saltzman E, Pieper CF, Fielding RA, Schwartz AV, Ravussin E, Redman LM; CALERIE-2 Study Group. Body-composition changes in the Comprehensive Assessment of Long-term Effects of Reducing Intake of Energy (CALERIE)-2 study: a 2-y randomized controlled trial of calorie restriction in nonobese humans. Am J Clin Nutr. 2017 Apr;105(4):913-927. doi: 10.3945/ajcn.116.137232. Epub 2017 Feb 22. PMID 28228420
- [Derived] Rochon J, Bhapkar M, Pieper CF, Kraus WE. Application of the Marginal Structural Model to Account for Suboptimal Adherence in a Randomized Controlled Trial. Contemp Clin Trials Commun. 2016 Dec 15;4:222-228. doi: 10.1016/j.conctc.2016.10.005. Epub 2016 Nov 3. PMID 27900372
- [Derived] Sparks LM, Redman LM, Conley KE, Harper ME, Yi F, Hodges A, Eroshkin A, Costford SR, Gabriel ME, Shook C, Cornnell HH, Ravussin E, Smith SR. Effects of 12 Months of Caloric Restriction on Muscle Mitochondrial Function in Healthy Individuals. J Clin Endocrinol Metab. 2017 Jan 1;102(1):111-121. doi: 10.1210/jc.2016-3211. PMID 27778643
- [Derived] Meydani SN, Das SK, Pieper CF, Lewis MR, Klein S, Dixit VD, Gupta AK, Villareal DT, Bhapkar M, Huang M, Fuss PJ, Roberts SB, Holloszy JO, Fontana L. Long-term moderate calorie restriction inhibits inflammation without impairing cell-mediated immunity: a randomized controlled trial in non-obese humans. Aging (Albany NY). 2016 Jul;8(7):1416-31. doi: 10.18632/aging.100994. PMID 27410480
- [Derived] Sanghvi A, Redman LM, Martin CK, Ravussin E, Hall KD. Validation of an inexpensive and accurate mathematical method to measure long-term changes in free-living energy intake. Am J Clin Nutr. 2015 Aug;102(2):353-8. doi: 10.3945/ajcn.115.111070. Epub 2015 Jun 3. PMID 26040640
- [Derived] Wong WW, Roberts SB, Racette SB, Das SK, Redman LM, Rochon J, Bhapkar MV, Clarke LL, Kraus WE. The doubly labeled water method produces highly reproducible longitudinal results in nutrition studies. J Nutr. 2014 May;144(5):777-83. doi: 10.3945/jn.113.187823. Epub 2014 Feb 12. PMID 24523488
- [Derived] Redman LM, Kraus WE, Bhapkar M, Das SK, Racette SB, Martin CK, Fontana L, Wong WW, Roberts SB, Ravussin E; CALERIE Study Group. Energy requirements in nonobese men and women: results from CALERIE. Am J Clin Nutr. 2014 Jan;99(1):71-8. doi: 10.3945/ajcn.113.065631. Epub 2013 Nov 20. PMID 24257721
- [Derived] Huffman KM, Redman LM, Landerman LR, Pieper CF, Stevens RD, Muehlbauer MJ, Wenner BR, Bain JR, Kraus VB, Newgard CB, Ravussin E, Kraus WE. Caloric restriction alters the metabolic response to a mixed-meal: results from a randomized, controlled trial. PLoS One. 2012;7(4):e28190. doi: 10.1371/journal.pone.0028190. Epub 2012 Apr 16. PMID 22523532
- See also: CALERIE website — https://calerie.duke.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 238 Participants were eligible, 18 participants withdrew prior to randomization, 220 participants were randomized to the study, and 2 participants withdrew prior to initiating the intervention.
Groups:
- Ad Libitum: Ad libitum energy intake
  Control: Participants continue their current diet for 24 months
Period: Overall Study
Arm/Group | Caloric Restriction (CR) | Ad Libitum
Started | 143 | 75
Completed | 117 | 71
Not Completed | 26 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caloric Restriction (CR) | Ad Libitum | Total
Number analyzed (Participants) | 143 | 75 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (7.3) | 38.1 (6.9) | 38.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 53 | 152
  Male | 44 | 22 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 111 | 57 | 168
  African-American | 15 | 11 | 26
  Other | 17 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Core Body Temperature, Baseline to 12 Months
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Caloric Restriction (CR) | Ad Libitum
Number analyzed (Participants) | 143 | 75
degrees Celsius | -0.05 (0.02) | -0.03 (0.02)
Statistical Analysis 1: Comparison: Caloric Restriction (CR) vs Ad Libitum; All analysis under intention-to-treat. All observations were included The primary analytic was a repeated measures analysis. The dependent variable was the change from baseline 12 & 14mos., with treatment, time, and the treatment × time interaction as independent variables. Site, sex, BMI stratum, and the baseline value of the outcome were included as covariates. The predicted mean changes ± standard errors are the adjusted values from the contrasts of the multiple timepoints; Test type: Other; p = 0.70, Mixed Models Analysis — Type I error was controlled using a hierarchical gatekeeping strategy; difference in mean change = 0.02, 95% CI 2-sided [-0.019 to 0.059], Standard Deviation 0.02

2. Primary Outcome: Change in Core Temperature, Baseline to 24 Months
Time Frame: Baseline to 24 months
Measure: Mean (Standard Deviation); unit: degrees Celsius
Groups:
- Prescribed 25% Caloric Restriction: 2 years of prescribed 25% Caloric Restriction
- Ad Libitum: Usual caloric intake
Arm/Group | Prescribed 25% Caloric Restriction | Ad Libitum
Number analyzed (Participants) | 143 | 75
degrees Celsius | -0.05 (0.02) | -0.02 (0.02)
Statistical Analysis 1: Comparison: Prescribed 25% Caloric Restriction vs Ad Libitum; Test type: Other; p = 0.84, Mixed Models Analysis; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.0092 to 0.069], Standard Error of Mean 0.02

3. Primary Outcome: Change in Resting Metabolic Rate (RMR) Corrected for Changes in Body Composition, Baseline to 12 Months
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: Kcal/day
Arm/Group | Caloric Restriction (CR) | Ad Libitum
Number analyzed (Participants) | 143 | 75
Kcal/day | -83 (10) | -1 (13)
Statistical Analysis 1: Comparison: Caloric Restriction (CR) vs Ad Libitum; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -82, 95% CI 2-sided [-103.8 to -60.2], Standard Error of Mean 11.12

4. Primary Outcome: Change in Resting Metabolic Rate (RMR) Corrected for Changes in Body Composition
Time Frame: Baseline, 24 months
Measure: Mean (Standard Deviation); unit: Kcal/day
Arm/Group | Caloric Restriction (CR) | Ad Libitum
Number analyzed (Participants) | 143 | 75
Kcal/day | -71 (12) | -7 (16)
Statistical Analysis 1: Comparison: Caloric Restriction (CR) vs Ad Libitum; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -64, 95% CI 2-sided [-90.5 to -37.5], Standard Deviation 13.5

5. Secondary Outcome: Change in Tumor Necrosis Factor-α (TNF-α), Baseline to 12 Months
Time Frame: change baseline to 12 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Caloric Restriction (CR) | Ad Libitum
Number analyzed (Participants) | 143 | 75
pg/mL | -0.30 (0.09) | -0.34 (0.12)
Statistical Analysis 1: Comparison: Caloric Restriction (CR) vs Ad Libitum; Test type: Other; p = 0.82, Mixed Models Analysis; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.16 to 0.23], Standard Error of Mean 0.10

6. Other Pre Specified Outcome: Change in Fat Mass
Description: Difference in change in Fat Mass between prescribed 25% Caloric Restriction (CR) and Ad Libitum (AL) at 12 and 24 months as measured by dual X-ray absorptiometry (DXA) using the Hologic 4500A, Delphi W or Discovery A, by a standardized protocol according to a standardized protocol. Fat Mass (FM) was determined for the whole body.
Time Frame: change 0 to 24 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Prescribed 25% Caloric Restriction | Ad Libitum
Number analyzed (Participants) | 143 | 75
kg | -6.1 (0.22) | -0.2 (0.28)
Statistical Analysis 1: Comparison: Prescribed 25% Caloric Restriction vs Ad Libitum; Difference in change in Fat Mass between prescribed 25% Caloric Restriction (CR) and Ad Libitum (AL) at 12 and 24 months as measured by dual X-ray absorptiometry (DXA) using the Hologic 4500A, Delphi W or Discovery A, by a standardized protocol according to a standardized protocol. Fat Mass (FM) and Fat Free Mass (FFM) were determined for the whole body; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -5.9, 95% CI 2-sided [-6.5 to -5.3], Standard Error of Mean 0.31

7. Other Pre Specified Outcome: Change in Fat Mass
Description: as for outcome 6
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Prescribed 25% Caloric Restriction | Ad Libitum
Number analyzed (Participants) | 143 | 75
Kg | -6.1 (0.22) | -0.3 (0.28)
Statistical Analysis 1: Comparison: Prescribed 25% Caloric Restriction vs Ad Libitum; Comparison of change in FM in 2 groups over at 24 mos, controlling for site, sex, BMI group, and baseline FM. A repeated measures Mixed Model was employed for the analysis. For any outcome, Type I error was controlled using a hierarchical gatekeeping strategy testing, first, the GroupXTime interaction, and, if non-significant, the main effects of these two factors. Bonferroni corrections were employed for non-significant effects. All tests were at p<0.05; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -5.9, 95% CI 2-sided [-6.4 to -5.3], Standard Error of Mean 0.26

ADVERSE EVENTS:
Time Frame: 0 to 24 months
Arm/Group | Caloric Restriction (CR) | Ad Libitum
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/143 | 7/75
Other Adverse Events (participants affected / at risk) | 136/143 | 72/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caloric Restriction (CR) (N=143) | Ad Libitum (N=75)
spontaneous miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
leiomyoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
intestinal abscess (Gastrointestinal disorders) | 0 (0) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
atrial septal defect (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caloric Restriction (CR) (N=143) | Ad Libitum (N=75)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 23 (43) | 8 (17)
dysmenorrhea (Reproductive system and breast disorders) | 30 (78) | 11 (31)
dizziness (General disorders) | 9 (48) | 10 (14)
diarrhea (Metabolism and nutrition disorders) | 20 (27) | 10 (16)
nasal congestion (General disorders) | 19 (28) | 5 (14)
constipation (General disorders) | 18 (44) | 5 (11)
toothache (General disorders) | 6 (21) | 5 (12)
muscle strain (Musculoskeletal and connective tissue disorders) | 3 (16) | 3 (4)
gastrointestinal virus (Infections and infestations) | 13 (16) | 5 (5)
pain (General disorders) | 12 (20) | 5 (10)
rash (General disorders) | 9 (9) | 1 (1)
urinary tract infection (Infections and infestations) | 4 (11) | 4 (6)
anemia (Blood and lymphatic system disorders) | 35 (99) | 17 (34)
Excessive bone loss (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — by BMD at lumbar spine, total hip and intertrochanter

LIMITATIONS AND CAVEATS:
1. The Caloric Restriction (CR) group fell short of achieving the 25% CR goal specified in the protocol.
2. The completion rates differed between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No